CLINICAL TRIAL: NCT05919745
Title: Patient Perception of Pain Following Extraction and Bone Graft Surgery With or Without Preemptive Ibuprofen: A Randomized Clinical Trial
Brief Title: Preemptive Ibuprofen Effects on Pain Perception Following Extraction and Bone Graft
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Vrisiis Kofina, Director, Advanced Education in Periodontics Program, Assistant Professor of Periodontics, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HR-4154
Record Dates: First submitted 2023-06-09; First posted 2023-06-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pain, Post Operative; Quality of Life
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen group or Test Group (Experimental): Subjects will be given ibuprofen 600mg tab 1h prior to surgery.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Acetaminophen
- Placebo group or Control group (Placebo Comparator): Subjects will be given a placebo tab 1h prior to surgery.
  Interventions: Drug: Placebo; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Preoperative delivery of ibuprofen per os.
  Other Names: Test
  Arms: Ibuprofen group or Test Group
Drug: Placebo — Preoperative delivery of placebo per os.
  Other Names: Control
  Arms: Placebo group or Control group
Drug: Acetaminophen — Both groups will be given rescue medication in the form of 1,000 mg tabs of acetaminophen every 6 hours per os as needed for pain (maximum allowed daily dose 4,000 mg per FDA) and will be allowed to receive ibuprofen or other analgesic medication as needed if pain is not controlled by acetaminophen alone. The subjects will receive the rescue medication pills at the end of the surgical appointment.
  Other Names: Rescue medication

SUMMARY:
The goal of this randomized clinical trial is to compare patient-reported pain and oral health-related quality of life during the first postoperative week following extraction and bone graft surgery in patients who received preemptive ibuprofen versus placebo. Participants will receive ibuprofen 600mg or placebo by mouth with water 1 hour prior to extraction and bone graft surgery.

The primary question it aims to answer is:

• Does preemptive ibuprofen have an effect on postoperative pain 1 hour following extraction and bone graft surgery compared to placebo?

Secondary questions are:

* Does preemptive ibuprofen have an effect on pain during the first 3 postoperative hours and 7 postoperative days following extraction and bone graft surgery compared to placebo?
* Does preemptive ibuprofen have an effect on oral health-related quality of life during the 7 postoperative days following extraction and bone graft surgery compared to placebo?

DETAILED DESCRIPTION:
The null hypothesis of this randomized clinical trial is that there is no difference in patient-reported pain and oral health-related quality of life during the first postoperative week following extraction and bone graft surgery between patients who received 600mg of preemptive ibuprofen versus placebo.

Participants will receive ibuprofen 600mg (test group) or placebo (control group) per os 1 hour prior to extraction and bone graft surgery. Researchers and patients will be blinded to the group assignment. Both groups will be given rescue medication in the form of 1,000 mg tabs of acetaminophen every 6 hours as needed for pain (maximum allowed daily dose 4,000 mg per FDA) and will be allowed to receive ibuprofen or other analgesic medication as needed if pain is not controlled by acetaminophen alone. The subjects will receive the rescue medication pills at the end of the surgical appointment.

Patient-reported pain will be collected by Visual Analogue Scale (VAS) before surgery, every hour for the first 3 postoperative hours and on postoperative days 1-7. VAS for patient-reported swelling will also be recorded at the same time points. Number of rescue medications will be recorded at the same postoperative time points. Oral health-related quality of life as expressed by Oral Health Impact Profile-14 (OHIP-14) questionnaire will be reported before surgery and on postoperative days 2, 5 and 7. Questionnaires on dental anxiety (Modified Dental Anxiety Scale), oral health literacy (Rapid estimate of Adult Literacy in Dentistry 30 Short Form), fear of pain (Fear of pain questionnaire-9) and pain catastrophizing (Pain catastrophizing scale) will be collected prior to surgery and will be evaluated as pain modifiers. Anticipated pain will be reported prior to surgery and questions on comparison between actual and anticipated pain and willingness to undergo a similar procedure again will be asked on days 1 and 7. Surgical and demographic data as well as medical history will be collected on the day of surgery. Clinical wound healing observations will be recorded on day 7.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years
* Good general health (controlled conditions)
* Fluent in English
* Treatment-planned for single site extraction and bone graft surgery

Exclusion criteria

* Pregnancy
* Site with active infection i.e purulence, abscess formation
* Patients experiencing pain pre-operatively
* Oral surgery in more than one site/quadrant in the same session
* Patients receiving surgery under sedation
* Patients with any contraindication for oral bone grafting surgery (e.g., on anticoagulants, medication-related osteonecrosis of the jaw, etc.)
* Patients experiencing acute or chronic oral pain due to conditions or previous interventions
* Patients with diseases or taking medications that affect hard and soft tissue wound healing such as poorly controlled diabetes, bisphosphonate use, corticosteroid use, chemotherapy, immunosuppressive therapy, etc.
* Current or chronic (≥4 weeks) use of anti-inflammatory, analgesic, corticosteroid or sedative medications in the past 6 months
* Health conditions that contraindicate the use of NSAIDs, such as stomach ulcers, bleeding disorders, renal disfunction, liver cirrhosis or acute liver disease, etc.
* Intake of medications that interact with NSAIDs or whose actions can be affected by NSAIDs, such as anticoagulant/antiplatelet medications, ACE inhibitors, diuretics, etc.
* Allergy to ibuprofen, acetaminophen and/or aspirin, and study materials (e.g., sutures, grafts, membranes?).
* Patients having 3 or more alcoholic beverages daily
* Patients who are planned to undergo heart surgery or had heart surgery less than 6 months prior
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in patient-reported postoperative pain between test and control group | 1 hour following extraction and bone graft surgery
  Visual Analogue Scale will be used to measure patient-reported pain. Its score range from 0-100 and the higher the score, the worse the reported pain is. Specifically, zero represents no pain and 100 represents the worst pain imaginable.

SECONDARY OUTCOMES:
Difference in patient-reported postoperative pain between test and control group | Postoperative hours 2 and 3, and postoperative days 1, 2, 3, 4, 5, 6 and 7 following extraction and bone graft surgery.
  Visual Analogue Scale will be used to measure patient-reported pain. Its score range from 0-100 and the higher the score, the worse the reported pain is. Specifically, zero represents no pain and 100 represents the worst pain imaginable.
Difference in Oral Health Impact Profile-14 between test and control group | Postoperative days 2, 5 and 7 following extraction and bone graft surgery
  Oral Health Impact Profile-14 is a validated widely used questionnaire that reliably measures oral health-related quality of life by recording patient perception of the impact of oral conditions on their well-being. Specifically, it consists of seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Its scores range from 0-56 and the higher the total score, the more impacted, i.e., worse, the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Vrisiis Kofina, DDS, MS, Principal Investigator — Marquette University
Locations (1):
- Marquette University School of Dentistry Graduate Periodontics Clinic, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No